CLINICAL TRIAL: NCT05562687
Title: Investigation of Association Between Single Nucleotide Polymorphisms in Genes of the Apelin/ APJ System (-1860T>C & G212A) and CAD Risk and Hypertension in Syrian Patients
Brief Title: Association Between Some Polymorphisms in Apelin/ Apelin Receptor Genes and Coronary Artery Disease in Syrian Patients
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDFP-Chemical-02-2022
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease; Hypertension
Keywords: Apelin; Apelin receptor (APJ); Coronary Artery Disease (CAD); Hypertension; apelin -1860T>C polymorphism; APJ G212A polymorphism
MeSH Terms: conditions — Coronary Artery Disease; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group: subjects who do not have any heart disease, hypertension, or other chronic &inflammatory diseases, and their coronary arteries are normal
- CAD group with essential hypertension: subjects who have stenosis (at least 70%) of one of the main coronary arteries or its branches and have high blood pressure
- CAD group without essential hypertension: subjects who have stenosis (at least 70%) of one of the main coronary arteries or its branches and have normal blood pressure
- Hypertension group without CAD: the subjects were characterized by the normal coronary artery and high blood pressure

SUMMARY:
The apelin-APJ signaling pathway has emerged as an important novel mediator of cardiovascular control and blood pressure homeostasis. Genetic variation in apelin and its receptors likely contributes to essential hypertension, in addition to a range of traditional risk factors. Thus, a study will be conducted on Syrian patients with hypertension and coronary artery disease to investigate some of the single polymorphisms in the apelin gene and its receptor that may be responsible for the development of these diseases, and to link the levels of this peptide and its receptor in the blood with these polymorphisms and the percentage of these diseases (as shown by many Modern Global Reference Studies).

DETAILED DESCRIPTION:
Blood levels of apelin and its receptor will be determined in patients and controls, and correlated with hypertension and coronary artery disease. And the allelic and genotypic frequencies of the G212A single polymorphism nucleotide of the apelin receptor gene and the -1860T>C single polymorphism nucleotide of the apelin gene in the study groups. And evaluation the functional role of A allele in hypertension. As well as investigating the association between: the genotypes of the apelin gene and the levels of apelin in the plasma, the genotypes of the apelin receptor gene and the levels of APJ in the plasma in the study groups. And link the polymorphism of the apelin gene with the polymorphism of the apelin receptor gene. And to determine the correlation between the presence of the studied SNPs and some traditional risk factors for coronary artery disease, which are age, hypertension, the onset age of hypertension, smoking, BMI, cholesterol and triglyceride levels in the blood, and family history of CAD.

ELIGIBILITY:
Inclusion Criteria:

* Control group: the subjects were characterized by no history of angina and other heart disease or hypertension, and do not have other chronic or inflammatory diseases.

They represent a normal resting ECG and normal exercise ECG stress testing. And the angiography showed the absence of any stenosis of the coronary arteries.

They were matched with CAD patients according to age, gender and ethnicity.

* CAD group with essential hypertension: the subjects were characterized by at least 70% stenosis in any coronary artery and high blood pressure (the average of three blood pressure readings was at least 140 mmHg systolic or 90 mmHg diastolic).
* CAD group without essential hypertension: the subjects were characterized by at least 70% stenosis in any coronary artery and normal blood pressure.
* Hypertension group without CAD: the subjects were characterized by the normal coronary artery and high blood pressure. And they were characterized by no history of angina and other heart disease or hypertension, and do not have other chronic or inflammatory diseases.

Exclusion Criteria:

* Individuals with valvular heart disease, cardiomyopathy, chronic kidney disease, diabetes, and inflammatory disease were excluded

Ages: 30 Years to 78 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Control group: subjects who do not have any heart disease, hypertension, or other chronic &inflammatory diseases, and their coronary arteries are normal.
  * CAD group with essential hypertension: subjects who have stenosis (at least 70%) of one of the main coronary arteries or its branches and have high blood pressure
  * CAD group without essential hypertension: subjects who have stenosis (at least 70%) of one of the main coronary arteries or its branches and have normal blood pressure
  * Hypertension group without CAD: the subjects were characterized by the normal coronary artery and high blood pressure.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Blood apelin concentrations | Collecting blood samples before angiography
  Blood samples will be obtained after a 10-h overnight fast before angiography and centrifuged at 1000 g for 10 min, then plasma specimens were stored at -80°C until analysis.
Blood apelin receptor (APJ) concentrations | Collecting blood samples before angiography
  Blood samples will be obtained after a 10-h overnight fast before angiography and centrifuged at 1000 g for 10 min, then plasma specimens were stored at -80°C until analysis
The allelic and genotypic frequencies of the -1860T>C single polymorphism nucleotides of the apelin genes | Collecting blood samples before angiography
  Genomic DNA will be extracted from peripheral blood sample, after that DNA will be stored in a deep freezer (-80°C) until the genetic analysis
The allelic and genotypic frequencies of the G212A single polymorphism nucleotides of the apelin receptor genes | Collecting blood samples before angiography
  Genomic DNA will be extracted from peripheral blood sample, after that DNA will be stored in a deep freezer (-80°C) until the genetic analysis.

SECONDARY OUTCOMES:
BMI | before angiography
  measurement of body weight and height will be recorded to calculate the body mass index
Measurement of blood pressure | before angiography
  Hypertension was diagnosed when the average of three blood pressure readings was at least 140 mmHg systolic or 90 mmHg diastolic, or in the event the individuals were taking antihypertensive medication
Plasma levels of triglycerides (TG) | Collecting blood samples before angiography
  Blood samples will be obtained after a 10-h overnight fast before angiography and centrifuged at 3000 g for 10 min, then plasma specimens were stored at -80°C until analysis
total cholesterol (TC) levels in plasma | Collecting blood samples before angiography
  Blood samples will be obtained after a 10-h overnight fast before angiography and centrifuged at 3000 g for 10 min, then plasma specimens were stored at -80°C until analysis
high-density lipoprotein cholesterol (HDL-C) levels in plasma | Collecting blood samples before angiography
  Blood samples will be obtained after a 10-h overnight fast before angiography and centrifuged at 3000 g for 10 min, then plasma specimens were stored at -80°C until analysis
low-density lipoprotein cholesterol (LDL-C) | Collecting blood samples before angiography
  Blood samples will be obtained after a 10-h overnight fast before angiography and centrifuged at 3000 g for 10 min, then plasma specimens were stored at -80°C until analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hussam Shebli, PhD, Study Director — Damascus university, ASPU Al-Sham Private University
Locations (1):
- Damascus University- Faculty of Pharmacy- Research and Graduate Studies Laboratory, Damascus, Syria

REFERENCES:
- [Background] Wang T, Liu C, Jia L, Ding J. The association between apelin polymorphisms and hypertension in China: A meta-analysis. J Renin Angiotensin Aldosterone Syst. 2019 Jan-Mar;20(1):1470320319827204. doi: 10.1177/1470320319827204. PMID 30755060
- [Background] Zhong JC, Zhang ZZ, Wang W, McKinnie SMK, Vederas JC, Oudit GY. Targeting the apelin pathway as a novel therapeutic approach for cardiovascular diseases. Biochim Biophys Acta Mol Basis Dis. 2017 Aug;1863(8):1942-1950. doi: 10.1016/j.bbadis.2016.11.007. Epub 2016 Nov 4. PMID 27825851
- [Background] Jin W, Su X, Xu M, Liu Y, Shi J, Lu L, Niu W. Interactive association of five candidate polymorphisms in Apelin/APJ pathway with coronary artery disease among Chinese hypertensive patients. PLoS One. 2012;7(12):e51123. doi: 10.1371/journal.pone.0051123. Epub 2012 Dec 3. PMID 23226564
- [Background] Falcone C, Bozzini S, Schirinzi S, Buzzi MP, Boiocchi C, Totaro R, Bondesan M, Pelissero G. APJ polymorphisms in coronary artery disease patients with and without hypertension. Mol Med Rep. 2012 Feb;5(2):321-5. doi: 10.3892/mmr.2011.685. Epub 2011 Nov 21. PMID 22109355
- [Background] Akcilar R, Yumun G, Bayat Z, Donbaloglu O, Erselcan K, Ece E, Kokdasgil H, Genc O. Characterization of the apelin -1860T>C polymorphism in Turkish coronary artery disease patients and healthy individuals. Int J Physiol Pathophysiol Pharmacol. 2015 Dec 25;7(4):165-71. eCollection 2015. PMID 27073592
- [Background] Huang F, Zhu P, Huang Q, Yuan Y, Lin F, Li Q. Associations between gene polymorphisms of the apelin-APJ system and the risk of hypertension. Blood Press. 2016 Aug;25(4):257-62. doi: 10.3109/08037051.2016.1156905. Epub 2016 Jun 24. PMID 27338090
- [Background] Nowzari Z, Masoumi M, Nazari-Robati M, Akbari H, Shahrokhi N, Asadikaram G. Association of polymorphisms of leptin, leptin receptor and apelin receptor genes with susceptibility to coronary artery disease and hypertension. Life Sci. 2018 Aug 15;207:166-171. doi: 10.1016/j.lfs.2018.06.007. Epub 2018 Jun 6. PMID 29883719
- [Background] Castan-Laurell I, Dray C, Valet P. The therapeutic potentials of apelin in obesity-associated diseases. Mol Cell Endocrinol. 2021 Jun 1;529:111278. doi: 10.1016/j.mce.2021.111278. Epub 2021 Apr 7. PMID 33838166